CLINICAL TRIAL: NCT04850664
Title: Development and Evaluation of Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) for Opioid Use Disorder
Brief Title: Computerized Chemosensory-Based Orbitofrontal Cortex (CBOT) for Opioid Use Disorder
Acronym: CBOT-OUD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evon Medics LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Howard University (Other); Family and Medical Counseling Service, Inc (Unknown); Maryland Treatment Centers @ ARTC (Unknown); Clinics of Dr. Edwin Chapman, MD, PC @ MHDG (Unknown)
Responsible Party: Principal Investigator, Evaristus Awele Nwulia, Chief Scientific Officer, Evon Medics LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CBOTDA049616; 2R44DA049616-02 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-04-20 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Opioid Use Disorder, Moderate; Opioid Use Disorder, Severe; Withdrawal Symptoms; Craving; Negative Affectivity
Keywords: Opioid Use Disorders; Buprenorphine Maintenance Treatment; Orbitofrontal cortex (OFC); CBOT; Relapse Prevention
MeSH Terms: conditions — Opioid-Related Disorders; Lymphoma, Follicular; Substance Withdrawal Syndrome | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Evon Medics will perform randomization of participants stratified by sex at site level. Site staff and participants will be blinded to treatment assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBOT + TAU (Experimental): CBOT consists of 40 cycles of olfactory stimulation and OFC training tasks, lasting ~45 minutes, once daily over 3 months. Treatment-as-usual (TAU) is standard dosing of buprenorphine (BUP) to a median dose of 24 mg (range 16-32 mg).
  Interventions: Drug: CBOT + TAU
- Sham + TAU (Sham Comparator): Sham is a CBOT device that uses artificially-scented compressed room air instead of olfactory stimulants and has no OFC cognitive tasks. Similar to the CBOT, sham will be used daily for 45 minutes. TAU is standard dosing of buprenorphine (BUP) to a median dose of 24 mg (range 16-32 mg).
  Interventions: Drug: Sham + TAU

INTERVENTIONS:
Drug: CBOT + TAU — The CBOT with proprietary odorant molecules is designed to stimulate olfactory neural activity over long periods of time. It is paired with OFC-dependent cognitive tasks.
  Other Names: plant based essential oils
  Arms: CBOT + TAU
Drug: Sham + TAU — Sham CBOT device uses artificially scented compressed room air instead of olfactory stimulants and has control cognitive tasks.
  Arms: Sham + TAU

SUMMARY:
Opioid Use Disorders (OUD) cause significant burden to individuals, families, and the society. Our product - Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT) - offers a cost-saving, home-based, user-friendly brain stimulation system that increased 6-month treatment retention of OUDs in a pilot study; and also, acutely reduced opioid withdrawal severity and negative affect during induction into opioid maintenance therapy. This study will establish its effectiveness in a broad category of OUD subjects at different stages of OUD care continuum.

DETAILED DESCRIPTION:
Evon Medics proposes to evaluate the effectiveness of Computerized Chemosensory-Based Orbitofrontal Cortex Training (CBOT), as an alternative strategy for relapse prevention in patients with Opioid Use (OUD) and other substance use disorders (SUD). This treatment leverages the overlap in brain regions that process smell and mediate decision making. The CBOT is portable and can be used at home. This clinical trial is being conducted to demonstrate its utility for home application by nontreatment seeking and treatment-seeking OUD populations, to engage in long-term, successful opioid recovery.

Key objectives of this project are to: (1) establish the effectiveness of CBOT for improved retention and relapse prevention in a large sample of OUD subjects; (2) establish its effectiveness for acute reduction of withdrawal severity and negative affect early in recovery; and (3) evaluate its safety, user-friendliness and acceptability. Accomplishment of these goals would lead to larger clinical trials for OUD and wider applications of CBOT in other addictive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 70years
* Diagnosis of current moderate or severe OUD in the past 6 months, including the past one month
* Willing to receive study interventions and buprenorphine during the study
* Do not meet criteria for current moderate or severe use of other substance use disorders (except nicotine use disorder)
* Diagnosis of Major Depressive Disorder, Anxiety disorders, and Post-traumatic Stress disorders will be included as long as the symptoms are stable, no suicidal ideas or plans and there are no recent changes in treatment of these conditions in the last 6 weeks prior to enrollment
* No intranasal disease
* Willing to participate by signing the informed consent form and
* Have a place to stay when receiving the intervention.

Exclusion Criteria:

* Any significant neurologic disease such as stroke, dementia, meningitis, neurosyphilis, cerebral palsy, encephalitis, epilepsy or seizures
* Mental retardation
* Schizophrenia or bipolar disorders
* Experiencing current suicide ideas or plans
* Any unstable medical condition such as uncontrolled hypertension, uncontrolled diabetes, and liver cirrhosis, as determined by site PI
* History of severe traumatic nose injury that affects ability to smell, as determined by site PI
* Allergies or intolerance to aromas from plant essential oils (e.g. orange and lemon)
* Breastfeeding or Pregnancy test positive.
* On parole or probation mandated to receive treatment for OUD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month buprenorphine maintenance treatment (BMT) retention | 2 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 4 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 6 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 8 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 10 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 12 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 14 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 16 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 18 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 20 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 22 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 24 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 26 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 28 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 30 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 32 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 34 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
6-month buprenorphine maintenance treatment (BMT) retention | 36 weeks after baseline
  6-month BMT retention is defined as missing two consecutive clinic visits after completing the first two weeks of BMT treatment, to allow for BUP dose stabilization.
  Ascertainment of retention is simply by tracking clinic visits and electronic record of the health visit.
Change from Screening in Subjective Opiate Withdrawal Scale (SOWS) at week | Screening to Week 12 Treatment
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely), and takes less than 10 minutes to complete.
Change from Screening in Subjective Opiate Withdrawal Scale (SOWS) at Week 24 | Screening to Week 24
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely), and takes less than 10 minutes to complete.
Change from Screening in Opioid Craving Scale (OCS) at Week 12 severity rating measures over 1 month | Screening visit to Week 12
  he Opioid Craving Scale, a modification of the Cocaine Craving Scale was used to measure opioid craving.
Change from Screening in Opioid Craving Scale (OCS) at Week 24 severity rating measures over 1 month | Screening visit to Week 24
  he Opioid Craving Scale, a modification of the Cocaine Craving Scale was used to measure opioid craving.
Change from Screening in negative affect severity in the PANAS | Screening visit to Week 12
  The Positive and Negative Affect Schedule (PANAS) is the most widely and frequently used scale to assess positive and negative affect.
Change from Screening in negative affect severity in the PANAS | Screening visit to Week 24
  The Positive and Negative Affect Schedule (PANAS) is the most widely and frequently used scale to assess positive and negative affect.

SECONDARY OUTCOMES:
Opioid Relapse | Screening visit to Week 12
  Relapse is defined as presence of self-reported repeated (i.e. 2 or more) use after the first two weeks for stabilization of buprenorphine dose, and/or presence of positive urine drug test for opiates. Ascertainment of opioid relapse is through: (a) Survey question administered 2-weekly, inquiring how days in the past did the subject use heroin, prescription opiates and/or other drugs; the dates of drug use; and the quantity (or dose) of drugs used; and (b) Biochemical verification of drug use, through urine samples will be collected and tested every two weeks.
Pre-Intervention changes in SOWS from Screening at Week 2 | Screening visit to Week 2
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Post-Intervention changes in SOWS from Week 12 at Week 13 | Week 12 to Week 13
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely).
Pre-Intervention changes in OCS from Screening to Week 2 | Screening visit to Week 2
  a modification of the Cocaine Craving Scale was used to measure opioid craving.
Post-Intervention changes in OCS from Week 12 to Week 13 | Week 12 to Week 13
  a modification of the Cocaine Craving Scale was used to measure opioid craving.
Pre-Intervention changes in PANAS negative affect from Screening visit to Week 2 | Screening visit to Week 2
  The Positive and Negative Affect Schedule (PANAS) is the most widely and frequently used scale to assess positive and negative affect.
Post-Intervention changes in PANAS negative affect from Week 12 at Week 13 | Week 12 to Week 13
  The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely). The Positive and Negative Affect Schedule (PANAS) is the most widely and frequently used scale to assess positive and negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Evaristus A Nwulia, MD, Principal Investigator — Evon Medics LLC; Tanya Alim, MD, Principal Investigator — Howard University; Mark Johnson, MD, Principal Investigator — Howard University; Marc Fishman, MD, Principal Investigator — Maryland Treatment Centers; Michael Serlin, MD, Principal Investigator — Family and Medical Counseling Service, Inc; Edwin Chapman, MD, Principal Investigator — Clinics of Dr. Edwin C. Chapman, MD, PC @ MHDG
Locations (4):
- United States (4):
  - Clinics of Dr. Edwin Chapman @ MHDG, Washington D.C., District of Columbia
  - Family and Medical Counseling Service, Inc, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Maryland Treatment Centers @ Avery Road Treatment Center, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson C, Rai N, McLean CK, Hipolito MMS, Hamilton FT, Kapetanovic S, Nwulia EA. Overlapping Risky Decision-Making and Olfactory Processing Ability in HIV-Infected Individuals. Clin Exp Psychol. 2017 Sep;3(3):160. doi: 10.4172/2471-2701.1000160. Epub 2017 Aug 15. PMID 29057388
- [Background] Volkow ND, Fowler JS. Addiction, a disease of compulsion and drive: involvement of the orbitofrontal cortex. Cereb Cortex. 2000 Mar;10(3):318-25. doi: 10.1093/cercor/10.3.318. PMID 10731226
- [Background] Lucantonio F, Takahashi YK, Hoffman AF, Chang CY, Bali-Chaudhary S, Shaham Y, Lupica CR, Schoenbaum G. Orbitofrontal activation restores insight lost after cocaine use. Nat Neurosci. 2014 Aug;17(8):1092-9. doi: 10.1038/nn.3763. Epub 2014 Jul 20. PMID 25042581
- [Background] Temple DM. Isolation techniques for pharmacologically active substances (animal). Annu Rev Pharmacol. 1969;9:407-18. doi: 10.1146/annurev.pa.09.040169.002203. No abstract available. PMID 4894805
- [Background] Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB. Effects of olfactory training in patients with olfactory loss. Laryngoscope. 2009 Mar;119(3):496-9. doi: 10.1002/lary.20101. PMID 19235739